CLINICAL TRIAL: NCT06399354
Title: The Effect of Medium-chain Fatty Acids on Cardiac Function
Acronym: MediHeart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Bente Kiens, Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MediHeart
Record Dates: First submitted 2024-04-09; First posted 2024-05-03 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Nutrition, Healthy; Heart Failure
Keywords: MCT; Glucose homeostase; ketogenese
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: A parallel, cross-over study in participants with heart failure and in a healthy age- and BMI-matched participants with normal heart function as control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meal test in patients (Experimental): Effect of medium-chain fatty acids on heart function measured by cardiac magnetic resonance imaging (CMR) in individuals with heart failure.
  Interventions: Dietary Supplement: acute intake of medium-chain fatty acids or long-chain fatty acids in patients
- Meal test in healthy individuals (Experimental): Acute intake of a meal comprising either MCT of LCT in healthy individuals and the effects onheart function.
  Interventions: Dietary Supplement: Acute intake of medium-chain fatty acids or long-chain fatty acids in healthy individuals

INTERVENTIONS:
Dietary Supplement: acute intake of medium-chain fatty acids or long-chain fatty acids in patients — The intake of an oil comprising of either medium -chain fatty acids or long-chail fatty acids
  Arms: Meal test in patients
Dietary Supplement: Acute intake of medium-chain fatty acids or long-chain fatty acids in healthy individuals — Acute intake of MCT and LCT in healthy individuals in a cross-over design
  Arms: Meal test in healthy individuals

SUMMARY:
The effect of an acute intake of medium-chain fatty acids on heart function measured by cardiac magnetic resonance imaging (CMR) will be measured in individuals with heart failure with reduced ejection fraction (HFrEF) and in matched healthy controls with normal heart function. This aim will be investigated in a cross-over study including two visits: acute intake of medium-chain fatty acid or long-chain fatty acid as control. In addition, the effect of acute medium-chain fatty acid compared with long-chain fatty acid intake on whole-body lipid and glucose metabolism will be investigated..

The hypothesis is that acute consumption of medium-chain fatty acid will improve cardiac function in patients with heart failure.

DETAILED DESCRIPTION:
The study will be conducted as a block-randomized cross-over study in participants with heart failure (HFrEF) (n=10) and in healthy age- and BMI-matched participants with normal heart function (n=13) as control group. The participants will undergo two experimental days separated by a two to four weeks wash-out period. At the test days, participants will consume cocoa milk added 0.5g/kg body weight of medium-chain fatty acid oil or long-chain fatty acid oil as control. Two days prior to metabolic testing, participants will consume a controlled diet. The controlled diet will be handed out to the participant.

Initially, potential participants are invited to an information meeting and after informed consent a screening is performed. Following inclusion, one of two identical test days are conducted consuming either medium-chain fatty acids or long-chain fatty acids in a randomized order. The participants will arrive after a 4 h period with no intake of food and drinks except water, and by passive transport (train, bus or car). After 30 min of rest in the supine position, venflon catheters are inserted into the right and left antecubital vein. After insertion of the catheters, fasting venous blood samples are drawn (20 ml in total) from one of the catheters for analysis of ketones, glucose, insulin, C-peptide, fatty acids, triacylglycerol, lipidomics and concentration of hepatokines. ECG monitoring is initiated. Thereafter, the first basal CMR will be performed.

After the basal blood sampling and scanning, the participants consume the cocoa-drink with 60g medium-chain fatty acid or 60g long-chain fatty acid and remains resting for the following 4 hours. Venous blood samples (15 ml) are obtained at 0, 30, 60, 80 and 135 min In total, up to 110 ml blood is obtained during the test day. At 90 min, the CMR will be repeated. At the end of the test day, the participant is served a meal. The duration of the test day is 4 hours. After a wash-out period of 2-4 weeks the test day will be repeated with consumption of the other fatty acid type.

ELIGIBILITY:
Inclusion Criteria for patients:

* Heart failure with reduced ejection fraction; I. Left ventricular ejection fraction ≤45% and optimal, stable HFrEF treatment according to guidelines II. Functional classification New York Heart Association class II-III.
* No uncorrected cardiac valvular disease
* No signs or symptoms of myocardial infarction within the previous 3 months
* No permanent of persistent arterial fibrillation.

For controls:

• No use of medications with influence on heart function

Exclusion Criteria: For all participants:

* Diabetes, kidney or liver disease.
* Contraindications to CMR, e.g., abdominal height exceed limitations of the MR- scanner, pacemaker, stent, neurostimulator, or other electronic device implanted, implanted metal devices, severe claustrophobia, or physiological diseases
* Pregnant, lactating or planning to become pregnant within the study period
* To ensure safety, no gadobutrol contrast can be administrered to participants with severe reduced kidney function, indicated by glomerular filtration rate (eGFR) < 30 ml/min/1.73m2, accessed from the obtained screening blood sample or from the Patient Record. In such cases, potential participants will be excluded from the study.
* Blood donation during and < 3 month prior to study
* Simultaneous participation in other clinical trials
* Inability, physically or mentally, to comply with the procedure required by the study protocol ad evaluated by the primary investigator, study manager or clinical responsible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Heart function | 0-5 weeks
  To investigate the effect of acute medium-chain fatty acids intake on heart function assessed by cardiac output (l/min) measured by cardiac magnetic resonance imaging (CMR) in individuals with heart failure with reduced ejection fraction (HFrEF) and in matched healthy controls with normal heart function.

SECONDARY OUTCOMES:
Measure of Ketones | 0-5 weeks
  Measure the effects of acute medium-chain fatty acid intake on plasma ketone concentration ( in mmol/l) as compared with long-chain fatty acid intake in individuals with and without heart failure.
Plasma Glucose | 0-5 weeks
  measure of plasma glucose concentration (in mmol/l) after the intake of medium-chain fatty acids as compared with the intake of long-chain fatty acids in individuals with and without heart failure
Measure of plasma lipids | 0-5 weeks
  measure of plasma triacylglycerol content in mmol/l after the intake of medium-chain fatty acids as compared with the intake of long-chain fatty acids in individuals with and without heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Bente Kiens, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark